CLINICAL TRIAL: NCT02214004
Title: A Phase II Trial of Preoperative HER2 Targeting and Endocrine Therapy in Postmenopausal Women With HER2 and HR Positive Breast Cancer
Brief Title: Neoadjuvant Trastuzumab and Letrozole for Postmenopausal Women
Acronym: HERAKLES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Seoul National University Hospital (Other); Severance Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERAKLES
Record Dates: First submitted 2014-08-05; First posted 2014-08-12 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; HER2; ER; Postmenopausal; Trastuzumab; Letrozole; Neoadjuvant endocrine treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab and Letrozole (Experimental): - Concurrently initiate two drugs on Day 1 of Cycle 1
  Interventions: Drug: Trastuzumab; Drug: Letrozole

INTERVENTIONS:
Drug: Trastuzumab — - Eight times IV administration of trastuzumab per 3 weeks
  * Trastuzumab 8mg/kg on Day 1 of Cycle 1
  * Trastuzumab 6mg/kg from Day 1 of Cycle 2 to Day 1 of Cycle 8
  Other Names: Herceptin
Drug: Letrozole — - Daily letrozole 2.5 mg/day for 24 weeks
  Other Names: Femara

SUMMARY:
The purpose of this study is to evaluate whether trastuzumab and letrozole are effective and safe in the preoperative treatment for postmenopausal patients with hormone receptor-positive and HER2-positive breast cancer.

DETAILED DESCRIPTION:
Eligibility criteria

* Ages Eligible for Study: ≥ 20 years
* Invasive cancer (clinical stage IB-IIIB)
* Measurable tumor larger than 1cm
* ECOG status 0 or 1
* Postmenopausal women

  * Age ≥55 years and amenorrhea
  * Age <55 years and amenorrhea for ≥12 months with FSH >30 mIU/ml
* HER2 positive tumor

  * 3 positive on IHC
  * 2 positive on IHC with HER2 gene amplification on FISH or SISH using a single-probe or dual-probe
* Estrogen receptor positive tumor

  * Positive ER expression with Allred score more than PS3/TS8 or modified Allred score more than PS4/TS7
* Eligible cardiac function

  * Normal heard evaluated by ECG

    * Consider clinically non-significant arrythmia and ischemic change as normal
  * LVEF ≥ 55% measured by ECHO or MUGA scan

Outcome measures

* Primary End-point

  * The rate of pathologic complete response (pCR)

    * No residual invasive cancer in breast
* Secondary End-point

  * Clinical Response Rate
  * Safety profiles for the preoperative use of concurrent trastuzumab and letrozole
  * The rate of breast conservative surgery
  * Total pathologic complete response (tpCR)

    * No residual invasive cancer in breast and ipsilateral axilla
  * Analysis of biomarkers based on baseline specimen and residual tumor
* Ki67 expression
* cDNA microarray: gene expression profiling
* Association between clinical response rate and circulating tumor cells (CTCs)

  * CTCs are measured by CytoGen (SEOUL, KOREA)"

ELIGIBILITY:
Inclusion Criteria:

* Invasive cancer (clinical stage IB-IIIC)
* Measurable tumor larger than 1cm
* ECOG status 0 or 1
* Postmenopausal women

  * Age ≥55 years and amenorrhea
  * Age <55 years and amenorrhea for ≥12 months with FSH >30 mIU/ml
* HER2 positive tumor

  * 3 positive on IHC
  * 2 positive on IHC with HER2 gene amplification on FISH or SISH using a single-probe or dual-probe
* Estrogen receptor positive tumor

  * Positive ER expression with Allred score more than PS3/TS8 or modified Allred score more than PS4/TS7
* Eligible cardiac function

  * Normal heard evaluated by ECG

    * Consider clinically non-significant arrythmia and ischemic change as normal
  * LVEF ≥ 55% measured by ECHO or MUGA scan

Exclusion Criteria:

* Inflammatory breast cancer
* Bilateral breast cancer
* Patients with previous breast cancer history
* Patients with previous breast cancer treatment: Generally include hormone therapy, chemotherapy, and radiotherapy)
* Patients having uncontrolled heart problems

  * Ischemic heart disease within 6 months
  * Congestive heart failure more than NYHA class II
  * Unstable angina
  * Clinically significant pericarditis
  * Amyloid heart disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The rate of pathologic complete response | At time of surgery
  No residual invasive cancer in breast regardless of axilla

SECONDARY OUTCOMES:
Clinical Response Rate | At time of surgery
  Clinical response includes complete response, partial response and stable disease.
Safety profiles for the preoperative use of concurrent trastuzumab and letrozole | Up to 3 months after surgery
  Toxicity according to CTCAE protocol from the initiated day to 3 months after surgery
The rate of breast conservative surgery | Up to 3 weeks after surgery
  The rate of breast conservative surgery among the patients receiving surgery
Total pathologic complete response (tpCR) | At time of surgery
  No residual invasive cancer in breast and ipsilateral axilla
Analysis of biomarkers based on baseline specimen and residual tumor | Baseline and at time of surgery
  * Ki67 expression
  * cDNA microarray: gene expression profiling
Association between clinical response rate and circulating tumor cells (CTCs) | Baseline and at time of surgery
  Association between clinical response rate and circulating tumor cells (CTCs)
  : CTCs are measured by CytoGen (SEOUL, KOREA)"

CONTACTS AND LOCATIONS:
Overall Officials: Joon Jeong, M.D.,Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (14):
- South Korea (14):
  - Hallym University Sacred Heart Hospital, Anyang
  - Inje University Pusan Paik Hospital, Busan
  - Dankook University Hospital, Cheonan
  - Ilsan Paik Hospital, Goyang
  - National Cancer Center, Goyang
  - Gangnam Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea Institute of Radiological and Medical Sciences, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: Undecided